CLINICAL TRIAL: NCT06983106
Title: Value of Automatically Segmented Three-Dimensional(3D) Volumetric Body Composition in Predicting the Pathological Grading and Prognosis of Gastroenteropancreatic Neuroendocrine Neoplasms: A Multicenter Study
Brief Title: Correlation Between Body Composition and Pathologic Grade/Prognosis in GEP-NENs: A Retrospective Study
Acronym: GEP-NENs
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhen Li, Professor, Tongji Hospital
Other Study IDs: TJ-IRB202411010
Record Dates: First submitted 2025-04-21; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: body composition calculate — The goal of this observational study is to learn about the value of body composition as predictors of pathological grading and prognosis in patients with gastroenteropancreatic neuroendocrine neoplasms. The volume of abdominal skeletal muscle and fat tissue is calculated based on CT scans at diagnosis.

SUMMARY:
The goal of this observational study is to learn about the value of body composition as predictors of pathological grading and prognosis in patients with gastroenteropancreatic neuroendocrine neoplasms.

The main question it aims to answer is: Does body composition affect the pathological grading and prognosis of patients with gastroenteropancreatic neuroendocrine tumors? Participants with gastroenteropancreatic neuroendocrine neoplasms will answer questions about their physical condition during follow-up visits.

DETAILED DESCRIPTION:
Objectives To explore the value of body composition parameters (BCPs) as predictors of pathological grading, prognosis in patients with gastroenteropancreatic neuroendocrine neoplasms (GEP-NENs).

Methods This retrospective multicenter analysis enrolled GEP-NENs patients pathologically confirmed from three institutions between 2015 and 2024. The volume of skeletal muscle and abdominal fat tissue was calculated based on CT scans at diagnosis. Univariate and multivariate logistic regression analyses were used to identify the relationships between BCPs and the pathological grade. The Kaplan-Meier method, along with the log-rank test, was employed for survival analysis. Independent prognostic factors were identified through uni- and multivariable Cox regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of GEP-NENs via histopathology with a WHO grading
* Available enhanced CT scans that included full abdominal imaging before surgery or biopsy

Exclusion Criteria:

* Therapeutic interventions before surgery or biopsy
* Poor image quality or incomplete CT images of the whole abdomen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective multi-center study involved three separate medical centers. Data from April 2015 to April 2024 were obtained from the respective hospital information systems, with CT scan images retrieved from the Picture Archiving and Communication System. Patients were included based on the following criteria: (1) a confirmed diagnosis of GEP-NENs via histopathology with a WHO grading; (2) available enhanced CT scans that included full abdominal imaging before surgery or biopsy. The exclusion criteria were: (1) therapeutic interventions before surgery or biopsy; (2) poor image quality or incomplete CT images of the whole abdomen. The WHO grading was derived from the postoperative pathology reports, which were meticulously reviewed and certified by experienced senior pathologists.
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
Correlation between CT-measured abdominal fat index(cm3/m3) and pathological grade (WHO classification) in GEP-NENs | Preoperative contrast-enhanced CT performed within one month before surgery
  Quantify abdominal visceral fat index(cm3/m3) ,subcutaneous fat index(cm3/m3) and intermuscular fat index(cm3/m3) using preoperative contrast-enhanced CT, and analyze their Pearson correlation coefficient with pathological grade (WHO classification: G1, G2, G3).

SECONDARY OUTCOMES:
Correlation between CT-measured abdominal fat index(cm3/m3) and 10-year overall survival (days) in GEP-NENs | From baseline CT to 10-year follow-up or death
  Quantify abdominal visceral fat index(cm3/m3) ,subcutaneous fat index(cm3/m3) and intermuscular fat index(cm3/m3) via preoperative CT, and analyze its Spearman correlation with overall survival (days from diagnosis to death) and progression-free survival (days from diagnosis to progression) using adjusted Cox proportional hazards models.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Li, Dr, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT06983106/Prot_SAP_000.pdf